Official Title: ICU experience among family members of ICU patients

**NCT** #: NCT02940028

**Document Date**: May 28 2020

#### Protocol

Title: ICU experience among Family Members of ICU Patients

**Location of Research:** Intermountain Medical Center

**Principal Investigator:** Ramona O. Hopkins, PhD

Sponsor: Intermountain Research and Medical Foundation

Study Team: Samuel M. Brown, MD

Jorie Butler, PhD Ellie Hirshberg, MD Sarah Beesley, MD James Orme, MD Tom Oniki, PhD Danielle Groat, PhD

#### **Purpose of the Study:**

The purpose of this study is to investigate whether an expressive writing intervention increases post-traumatic growth (PTG) in family members of patients admitted to the ICU with a serious illness and explore the association between coping phenotypes and PTG. PTG will be compared between the intervention group receiving the expressive writing intervention and the control group (non-expressive or fact-based writing). The primary outcome will be PTG at 12 weeks, with secondary outcomes of depression, anxiety and posttraumatic stress disorder (PTSD) at follow up.

# **Hypothesis/Research Questions:**

In two hypotheses evaluated in two specific aims, we will investigate whether an expressive writing intervention increases PTG in family members of patients admitted to the ICU with a serious illness and explore the association between coping phenotypes and PTG. PTG will be compared between the intervention group receiving the expressive writing intervention and the control group (non-expressive or fact-based writing). The primary outcome will be PTG at 16 weeks, with secondary outcomes of depression, anxiety and PTSD at follow up.

# Specific Aim 1: Examine the association between participating in an expressive writing intervention and development of post-traumatic growth.

<u>Primary outcome</u>: Post-Traumatic Growth Inventory at 4 months <u>Secondary outcomes</u>: Impact of Events Scale-Revised (IESR), Hospital Anxiety and Depression Inventory (HADS) at 4 months

**Hypothesis 1a:** Participants in the intervention group will have higher levels of post-traumatic growth at follow-up than participants in the control group.

**Hypothesis 1b:** Participants in the intervention group will have lower PTSD, depression, and anxiety scores at 4 months.

**Specific Aim 2:** Explore whether individual coping phenotypes predict PTG. Predictors for consideration include acute perceived stress (Perceived Stress Scale-4 [PSS-4], personality characteristics (Big Five Inventory [BFI]) coping ability (Brief COPE), social relationship quality (Social Relationship Inventory (SRI abbreviated), measures of disability in activities of daily living and instrumental activities of daily living caregiver burden (Groningen Activity Restriction [GARS] Scale), patient age and severity of illness (APACHE score).

**Hypothesis 2a:** ICU families coping phenotypes (stress, personality characteristics, and coping) will be associated with PTG.

**Hypothesis 2b:** Other variables related to the ICU (APACHE IV score, age, sex, ethnicity, whether the patient dies before follow-up) and post-ICU (care giver burden) experience will be associated with PTG at 3 mos.

# **Background and Significance:**

# Post-ICU psychological distress is common and important

The intensive care unit (ICU) is a stressful and challenging place for patients and their families, who must navigate illness and its associated discomforts as well as complex decision making in an environment characterized by tremendous uncertainty<sup>1-3</sup>. Negative emotions including stress, fear, anger, and fatigue are extremely common during an ICU admission<sup>4,5</sup>. Many family members experience anxiety, depression, and posttraumatic stress disorder (PTSD) during and after the ICU experience that persists years after their loved one is discharged from the ICU<sup>3,6-8</sup>.

During an ICU stay, it is common for patients to be too ill to participate in decision making in the ICU<sup>9</sup> – and medical decision making will generally be made by the family members designated surrogate decision makers<sup>7</sup>. Surrogate medical decision making may be intense and stressful and may contribute to development of anxiety, depression and posttraumatic stress disorder (PTSD) in family members <sup>3</sup>.

Persistent psychological distress after ICU admission is part of a recognized syndrome called post-intensive care syndrome-Family (PICS-F)<sup>10</sup>. The reasons for PICS-F in response to the emotional trauma of the ICU are multifactorial, and include pre-existing risk factors, failures to meet informational needs, threat of death or serious disability, and decision-related stress, given the heavy psychological burden associated with decision making about matters of life and death<sup>1,3</sup>. Traumatic experiences, however, can also result in positive psychological outcomes – including better relationships, improvements in spiritual well-being, greater self-efficacy, and personal development. Such positive post-trauma outcomes are known as post-traumatic growth (PTG)<sup>11</sup> and may represent an alternative to the PTSD and anxiety that have come to the hallmark of PICS-F.

# Post-traumatic growth

Post-traumatic growth is a positive change in a person's sense of self that is part of a complex narrative or personal life story that occurs after a difficult life experience. An individuals' world view with the accompanying goals, beliefs, and habits of managing emotional feelings and stress can be shaken by traumatic experiences and then, over time, are rebuilt into a new positive view of the self and life<sup>11-13</sup>. Post-traumatic growth (PTG) has been observed in response to a wide variety of traumatic experiences including medical illnesses (chronic illness, cancer, AIDS), military combat, man-made disasters (e.g., shootings) and natural disasters (e.g., tornadoes)<sup>14,15</sup>. Patterns of PTG vary based on aspects of the trauma and the individual's characteristics. Some evidence suggests that the traumatic events associated with the greatest PTG represent intermediate levels of harm. Personal characteristics associated with PTG, include openness, extraversion, agreeableness and conscientiousness alternatively neuroticism is associated with less PTG. Greater PTG is associated with -focused coping and cognitive processing of the traumatic event, involvement in religious activities and high levels of perceived social support<sup>15-17</sup>. Overall, some degree of emotional processing of the traumatic event must take place for PTG to occur,<sup>12</sup> and such processing is most likely to result in post-traumatic growth in a particular personal and social context.

Post traumatic growth takes time to emerge, with most positive changes occurring within 2 months after the trauma<sup>18</sup> while the level of PTG remains stable 3 to 8 years following the trauma<sup>19,20</sup>.

# **Potential Benefits of Expressive Writing**

Although PTG is a naturally occurring process, deliberate interventions can increase its likelihood. Some interventions are time-consuming and expensive – such as cognitive behavioral therapy. But, in some contexts, interventions centered on a specific type of journaling known as "expressive writing" have increased PTG. Semi-structured expressive writing was developed by James Pennebaker, Ph.D. as a structured technique for recording deep thoughts and feelings about a traumatic event in a structured setting <sup>21</sup>. Expressive writing facilitates coping with trauma by helping people process – emotionally and cognitively – a traumatic event. Participating in expressive writing – commonly three 20-minute sessions on three consecutive days – includes writing about emotions and thoughts associated with the traumatic event. Variations include providing participants with a journal and asking them to complete the writing at set times at home<sup>22</sup> or using an internet-based journal<sup>23</sup>. In many studies expressive writing interventions are associated with improved outcomes including fewer reports of physical symptoms, a reduction in PTSD and greater PTG<sup>22-24</sup>. In addition, expressive writing is associated with reduced healthcare utilization, fewer physical symptoms, and fewer PTSD symptoms on follow-up<sup>21,22,25</sup>.

Family members and patients enter the ICU with unique characteristics that may affect their risk for psychological distress<sup>26</sup>. In other trauma-exposed populations, individual attributes have been associated with development of PTSD<sup>26,27</sup>. Personalizing the experience of family members by offering post-ICU support strategies, such as writing interventions, may decrease psychological distress and improve positive outcomes and PTG<sup>11,28</sup>.

In prior work, we identified ICU family member coping phenotypes that would identify individual attributes, preferences, and vulnerabilities (personality dimensions, shared decision-making preferences, coping styles, and social support) that might be relevant to the experience of ICU surrogates<sup>29</sup>. We identified three copying phenotypes including adaptive copers, maladaptive copers, and disengaged copers. Coping phenotypes differed primarily on coping styles, personality, quality of their closest social relationship, and history of anxiety and depression.<sup>29</sup> Early work suggests that individuals in certain coping phenotypes may have different approaches to surrogate decision making and different satisfaction with the shared decision making during a simulated ICU experience. They may also have different probabilities of PTG.

# **Research Subjects:**

#### Inclusion Criteria:

Family members of ICU patients are eligible for the study. We will enroll **one** study participant per patient admitted to a study ICU (Shock Trauma or Respiratory ICU at Intermountain Medical Center) who meets the following inclusion criteria:

- Participant can be a family member of a patient admitted to a study ICU for >24 hours and >1
   of the following:
  - mechanical ventilation via endotracheal tube for ≥ 12 hours
  - non-invasive ventilation (CPAP, BiPAP) for > 4 hours in a 24-hour period provided for acute respiratory failure in an ICU (not for obstructive sleep apnea or other stable use)
  - high flow nasal cannula or face mask O2 with FiO2 ≥ 0.5 for ≥4 hours
  - use of vasopressors for shock of any etiology for >1 hour
- The priority for enrollment is outlined in the picture below.

#### Does the potential participant live with the patient? **PREFERRED ACCEPTED** If YES, then: If NO, then: 1. Do they have designated power of attorney? 1. Do they have designated power of attorney? 2. Are they the primary caretaker? 2. Are they the primary caretaker? 3. Are they the default surrogate?\* 3. Are they the default surrogate?\* MUST HAVE AT LEAST ONE OF THE ABOVE QUALIFICATIONS MUST HAVE AT LEAST ONE OF THE ABOVE QUALIFICATIONS \* A default surrogate can include (in order of preference): 2. Adult child 1. Spouse (unless divorced or legally separated OR if court 3. Parent 4. Sibling finds spouse acted in a manner 5. Grandparent that should preclude him/her 6. Grandchild from having a priority position)

- Both participant and ICU patient must be adult (age ≥18 years of age)
- Participant must be able to read, speak, and write in English
- Participant must be enrolled within 72 hours of the patient's meeting mechanical ventilation criteria.

Participants who live with the patient will be accorded higher priority than those who do not live with the patient because they are more likely to be involved as caregivers. The preference would be for the

participant to be the designated power of attorney; if there is no designated power of attorney living with the patient, then the primary informal caregiver (identified either by the patient or by the family) would be enrolled; if either of these is not available, the default surrogate (defined in figure 1) would be enrolled. If no one living with the patient meets these criteria, then family members and informal caregivers not living with the patient will be screened for the study. The preference would again be for first, the designated power of attorney, then a primary caregiver and a default surrogate. An informal caregiver provides care without reimbursement.

#### Participant Exclusion Criteria:

- Pregnant or breastfeeding females
- Prisoners
- Children (age <18 years of age)</li>
- Known history of PTSD, dementia, or schizophrenia. Presence of these illnesses will be per participant report of physician diagnosis and treatment
- If a patient has been transferred from another ICU after an ICU course greater than 24 hours, or if the patient has had a previous ICU or long-term acute care (LTAC) admission in the last 90 days, the family member or caregiver will be excluded.
- Patients admitted for hospice
- Participants who live more than 200 miles away or who have no specified domicile
- Non-English speaking

Because ICUs are sometimes used for simple monitoring of patients with low severity of illness and that experience is likely to be quite different from an admission for critical illness, we restrict to patients with at least a moderate severity of illness as judged by >48 hours of mechanical ventilation. We exclude participants who have underlying mental disease such as PTSD, dementia, and schizophrenia because these participants may process trauma-related information very differently from other participants. The intervention features expressive writing so understanding, speaking, and writing in English is critical as we will not have the capacity to conduct data analysis of the writing sample in other languages. We are most interested in subjects who have experienced acute stress at an identifiable time (during the ICU admission) thus family members who have already been in ICU or in other critical care environments may not be undergoing acute stress.

#### Recruitment:

Qualified study participants will be consented prior to commencing any research-related activity. These individuals will be approached in the patient's room or waiting room in the ICU or by telephone.

# Methods/Procedures: Baseline Assessment

Participants will be enrolled in the study if they meet study inclusion and no exclusion criteria and signed informed consent. Participants will be administered baseline questionnaires, randomly assigned to the intervention or control condition, participate in intervention or control writing condition at 4 weeks (range 2 to 8 weeks) after enrollment, and administered follow-up questionnaires at three months after the writing intervention (± 2 weeks) by telephone.

# Questionnaires

Participants will complete baseline questionnaires including<sup>32</sup>, PSS-4, BFI, Brief COPE, HADS and the IESR.

Table 1. Questionnaires administered at study enrollment

| Instrument | Measures | Scale | Scoring |
|---|---|---|---|
| Hospital Depression | Depression and anxiety | 14 items (7 each for | Scores of 8 or |
| and Anxiety Scale | | anxiety and | higher indicate |
| | | depression). Items | symptoms or |
| | | scored 0 to 3. Total | depression or |
| | | scores for each scale | anxiety. <sup>33</sup> |
| | | range from 0 to 21. | |
| Impact of Event Scale | Screens for PTSD | 22-item scale | A mean score of ≥ |
| Revised (IES-R) | | measuring intrusion, | 1.6 indicates PTSD |
| | | avoidance and | symptoms. <sup>34,35</sup> |
| | | hyperarousal; each | |
| | | item scored from 0-4 | |
| Perceived Stress Scale | Feelings of stress | 4 items with scores | Higher scores |
| | | that range from 0 to | indicate greater |
| | | 4 | stress. <sup>36,37</sup> |
| Brief COPE | Coping with stress | 14 dimensions with 2 | Higher scores |
| | | questions per | indicated greater |
| | | dimension | use of a given |
| | | | coping strategy. <sup>38</sup> |
| Social Relationship | Quality of Social Support | 3 dimensions of | Higher scores on |
| Inventory (abbreviated) | | relationship for the | each dimension |
| | | person closest to | indicate greater |
| | | the respondent, | helpfulness, upset, |
| | | helpfulness, upset, | and unpredictability. |
| | | and unpredictability | |
| | | rated from 1 (not at | |
| | | all) to 6 (extremely) | |
| Big Five Inventory | Personality dimensions: | 10 items | Higher scores |
| | openness to new experiences, | | indicate greater |
| | conscientiousness, extra | | degree of a specific |
| | version, agreeableness and | | personality |
| | neuroticism. | | characteristic. <sup>39</sup> |

# **Random Assignment and Intervention**

Random assignment to condition will be completed using random number generator. Participants will receive instructions for participating in the intervention.

The intervention will take place in person at 4 weeks ( $\pm$  2 to 8 weeks). Participants will participate in a semi-structured 20-minute expressive writing session in person or at home with instructions. For those in the experimental expressive writing condition, the instructions (adapted from Stanton & Danoff-Burg)<sup>24</sup> will be:

"What I would like you to write about for these three sessions are your deepest thoughts and feelings about your experience with your family member in the Intensive Care Unit (ICU). I realize that people with a loved one in the ICU experience a full range of emotions and thoughts, and I want you to focus on any and all of them. In your writing, I want you to really let go and explore your very deepest emotions and thoughts. You might think about all the various feelings and changes that you experienced before your loved one was hospitalized in the ICU, after the diagnosis that led them to the ICU, during treatment, and now. Whatever you choose to write, it is critical that you really focus on your deepest thoughts and feelings. Ideally, I would like you to focus on feelings, thoughts, or changes that you have not discussed in great detail with others-private feelings. You might also tie your thoughts and feelings about your experiences with having your loved one in the ICU to other parts of your life, i.e., your childhood, people you love (this loved one and others), who you are, or who you want to be. Again, the most important part of your writing is that you really focus on your deepest emotions and thoughts. The only rule we have is that you write continuously for the entire time. If you run out of things to say, just repeat what you have already written. Don't worry about grammar, spelling, or sentence structure. Don't worry about erasing or crossing things out. Just write."

Participants in the control condition will receive the following instructions:

"What I would like you to write about for these three sessions are all the facts about your experience with your family member in the Intensive Care Unit (ICU). We are not interested in your thoughts and emotions. Please do not include them. We are interested in all the facts about how your loved one came to the ICU and the facts about your experiences in the ICU with your loved one. The only rule we have is that you write continuously for the entire time. If you run out of things to say, just repeat what you have already written. Don't worry about grammar, spelling, or sentence structure. Don't worry about erasing or crossing things out. Just write."

Participants will write for 20 minutes for 3 sessions that will occur over a 2-hour period on the participation day (8 weeks after the hospitalization). Participants who are comfortable typing will type responses into a REDCap website via a tablet and keyboard which will measure the amount of time spent writing or at home on their computer and will email the writing sample to the study coordinator.

Participants who use handwriting will be observed by the project coordinator if in person. Instructions will be sent to the participant if completing the writing at home.

- a. Study coordinator will call the study participant to assess if they are willing and able to do the writing at home and set up a date and time for them to do the writing follow-up at home.
- b. Each participant will be sent a unique identifier (ex. 193JTA) that we will link to study ID and them they will be instructed use the code to identify their writing instead of their name.
- c. An instruction sheet will be emailed or sent to the participant via email or regular mail if writing long hand.
- d. The participants will be instructed to use the identifier in the subject line of email when they send the writing sample back to the study coordinator Mardee Merrill at <a href="Mardee.Merrill@imail.org">Mardee.Merrill@imail.org</a> or to Ramona Hopkins, PhD at <a href="Mona.Hopkins@imail.org">Mona.Hopkins@imail.org</a>.

e. If writing is done long-hand a self-addressed stamped envelope will be included to send back the writing to the study coordinator.

Manipulation checks include completion of the Essay Evaluation form in which participants will rate how personal, meaningful, and reflective of their feelings their essay is. Participants in the control condition should rate this very low in comparison to participants in experimental conditions. All participants who complete follow up will receive a gift card after completing the writing intervention.

# 4 Month Follow-up

Four months after the writing exercise, participants will be contacted to complete an instrument battery by telephone. Follow-up measures include IES-R, HADS, PSS-4, Groningen Activities Restriction Scale (GARS) for assessing impact of the traumatic event on functional and emotional health and Posttraumatic Growth Inventory (PTGI). Following participation participants will receive gift card payment in the mail.

| 4 Month Follow | <i>r</i> -up | | |
|---|---|---|---|
| Hospital<br>Depression<br>and Anxiety<br>Scale | depression and anxiety | 14 items (7 each for anxiety and depression). Items scored 0 to 3. Total | Scores of 8 or higher indicate symptoms or depression or anxiety. <sup>33</sup> |
| Impact of<br>Event Scale<br>Revised (IES-<br>R) | Screens for PTSD | 22-item scale measuring intrusion, avoidance and hyperarousal | A mean score of ≥ 1.6 indicates PTSD symptoms. 34,35 |
| Perceived<br>Stress Scale | Feelings of stress | 4 items with scores that range from 0 to 4 | Higher scores indicate greater stress. <sup>36,37</sup> |
| Brief COPE | Coping with stress | 14 dimensions<br>with 2<br>questions per<br>dimension | Higher scores indicated greater use of a given coping strategy. <sup>38</sup> |
| Post-<br>Traumatic<br>Growth<br>Inventory | Positive perceptions of change following a traumatic event | 21 items that<br>use a 6 point<br>Likert scale (0-<br>5) | Higher Scores Indicate greater PTG |
| Physical<br>Symptoms<br>Inventory – 13<br>Item Version | Examines physical symptoms experienced during previous 30 days adapted to include medical utilization | 13 items that<br>use a 5 point<br>Likert Scale (1-<br>5) | Higher scores indicate more symptoms on more days. |

| Groningen<br>Activity<br>Restriction<br>Scale (GARS) | Assess degree of restriction experienced due to providing care in 11 categories: caring for him/herself, caring for others, eating habits, shopping for him/herself, visiting friends, working on hobbies, sports and recreation, going to work, and maintaining friendship. Developed and used in ICU populations, 46-49 shopping for him/herself, visiting friends, working on hobbies, sports and recreation, going to work, and maintaining friendship. and used in ICU populations. 46-49 | 11 items scored from 1 to 4 | Scores range from 11 to 44 with higher scores indicating greater activity restriction. |
|---|---|---|---|
| Groningen<br>Activity<br>Restriction<br>Scale (GARS) | Assess degree of restriction experienced due to providing care in 11 categories: caring for him/herself, caring for others, eating habits, sleeping habits, doing household chores, going | 11 items scored from 1 to 4 | Scores range from 11 to 44 with higher scores indicating greater activity restriction. |
| Essay<br>Evaluation<br>Measure | Perception that essay was personal, meaningful and revealing of their emotions | Each item<br>Likert 0-6 total<br>range 0-18 | Higher scores indicate that participants found the essay personal and meaningful and revealing of their emotions (0-18) <sup>50</sup> |
| | Evaluation of essays not done with participant | | |

#### **Informed Consent:**

Study-designated Intermountain Healthcare employees (either the research coordinator(s) or the study investigator(s)) will obtain informed consent from the study participant. The study staff member obtaining consent will provide the participant with the current IRB-approved Informed Consent Form and will be available to answer any questions the participant may have. Individuals approached for consent will be given as much time as they require to consider enrollment in the study.

The ICU patient will not be approached or questioned. They are indirectly involved, as the study participant is defined by their relationship to the patient. Minimal information will be obtained about the patient from the medical record to allow assessment of the effects of acute severity of illness or length of stay. The ICU patient will not be consented as they are not the subject of the study and minimal information is collected regarding these individuals. We will ask for a waiver of informed consent to gather this data.

#### **Waiver of Informed Consent**

The ICU patients are not directly involved and will not be approached or questioned. Minimal information will be obtained about the patients. The ICU patients will not be consented as they are not the subject of the study and minimal information is collected regarding these individuals. We will ask for a waiver of informed consent to gather this data. We feel it is not necessary or appropriate to obtain consent from the ICU patients for these reasons.

Only the minimum PHI needed will be collected. We will only collect names, hospital ID number and dates necessary to determine hospital and length of ICU stay. The study data will be stored on secure computers and will be de-identified. We will protect confidentiality and privacy in a HIPAA- and Good Clinical Practice- compliant way. Subjects will be given an anonymous study ID. In addition to managing only non-identified data, we will also protect that data by storing it only on secure computers. The only data sharing will be with our collaborator Dr. Jorie Butler at the University of Utah. All other data sharing such as might be required for regulatory reasons or to comply with editorial requirements of scientific journals, will be deidentified.

#### Risks:

Based on prior research in psychology and in critical care, we anticipate that there will be only minimal risk to those participating in this research. Patients may experience some discomfort from answered survey questions and writing about their family members ICU experience. In our experience surveying many hundreds of patients and families during and after an ICU admission, this is very uncommon. Participants are always free to decline to answer any question or further participation. Breach of confidentiality is a potential risk, but the data will be appropriately safeguarded against inappropriate disclosure.

#### **Benefits:**

Data indicate that ICU admission results in adverse psychological outcome including depression, anxiety and posttraumatic stress disorder. If the intervention enhances PTG, we will be able to help family members of critically patients develop positive outcomes. Our ultimate goal is to understand, predict, and improve psychological outcomes (depression, anxiety and PTSD) in patients and their family members after ICU admission. This study may help future ICU patients and their family members by helping us to understand how PTG may affect psychological wellbeing for family of patients admitted to the ICU

## Impact on Intermountain

Intermountain Medical Center is a pioneer in the study of long-term outcomes after critical illness and patient- and family-centered intensive care. We plan to expand these investigations into a better understanding of the long-term outcomes and acute patient- and family-related experiences associated with an ICU admission more generally. This work will allow us to expand prior expertise and reputation in the field of long-term outcomes after critical illness and to establish Intermountain Medical Center as a leader in interventions during critical illness that improve long-term outcomes. We see this research project as a key way to further cement Intermountain's profound leadership in creating ICUs that are carefully attuned to the human side of serious illness.

# **Compensation:**

If participants decide to participate in the study, to compensate them for their time and effort, at the writing exercise visit, they will receive a \$50 gift card or be mailed a \$50 check. After the 4-month follow-up phone call, they will receive another \$50 gift card or be mailed a \$50 check. Thus, if they complete the study, they will receive a total of \$100 for the two visits.

#### **Data Collection:**

**Demographic Characteristics:** Participant age, sex, ethnicity, years of educational attainment, identification with religion (e.g., Buddhism, Christian, Muslims well as "Spiritual but not religious" or "other") were collected. The importance of religion was assessed using the following questions: (*How important is religion in your daily life?*) from (1) *not at all* to (4) *extremely* and religious service attendance (*How frequently do you attend religious services?*). History of anxiety and depression were assessed (e.g., *Do you have a personal history of anxiety?*), and whether they had ever received treatment by a physician or mental health provider.

This study requires the use of the following information:

- ICU Patient information (the only PHI required is the hospital ID number used to collect the non-PHI demographics and outcome information)
  - o Age (if the patient's age is greater than 89, it will be recorded as 89)
  - Sex
  - o Race
  - o Ethnicity
  - Primary ICU diagnosis
  - APACHE II score at admission
  - Prior ICU admissions in the last 5 years (per report from participant)
  - Mortality at 3 months (i.e., living or deceased per report from participant)
  - Hospital and ICU length of stay
  - Presence of mechanical ventilation
  - Baseline terminal illness (congestive heart failure, ESRD, liver failure, cancer)
- Study Participant information:
  - Age
  - o Sex
  - Race
  - Ethnicity
  - Religion (importance, affiliation, and degree of importance)
  - Employment status
  - Number of hours weekly spent with the patient (averaged over the last month) and whether the participant lives with the patient,
  - Highest level of education.
  - Limited medical history: diagnosed depression, anxiety, sleep disorder, obesity. 30,31
  - Psychiatric history of depression or anxiety
  - History of substance and alcohol abuse

The informed consent form describes the elements of PHI that will be used as a part of this study. All identifiable study information that is collected will be kept on computers owned and secured by Intermountain Healthcare. Any PHI collected for this study will be de-identified prior to disclosure to study collaborators outside of Intermountain Healthcare and only under authorization of current, valid data use agreements. The code used to de-identify these subjects will be retained by the Intermountain Healthcare Principal Investigator to allow re-identification of the subject should clarification of information be required. Identifiers of study participants will be maintained securely in order to report study results to participants, e.g., via newsletters.

We will randomize family members to receive either the PTG intervention and or non-intervention control group (control writing condition). The intervention group will participate in a brief expressive writing intervention. The control group will receive a control writing condition (fact-based writing) and complete the other study measures.

Descriptive statistics will be calculated for all demographic variables as well as all instruments (both at baseline and 4 month follow up). PTGI at 4 months (along with the secondary outcomes) will be compared between the intervention and control arms using Wilcoxon Rank Sum tests. Further, we will use linear regression to assess the relationship between expressive writing and PTGI at 4 months, adjusting for other relevant factors (i.e., participant demographics, (including age), patient demographics, illness severity of the patient, social support of the participant, caregiver burden, etc.).

# Sample Size:

Studies of post-traumatic growth using the PTGI have sample means ranging from 45-77 <sup>51 52-55</sup>. We hypothesize that participants in the intervention arm will have a higher PTGI at 4 months compared to those in the control arm. Based on previous studies, we assumed a mean (SD) PTGI at 4 months of 45 <sup>18</sup> in the control arm and 56 <sup>21</sup> in the intervention arm <sup>23,52,53</sup>. A power analysis based on the Wilcoxon Rank Sum test determined 102 patients are necessary to identify a significant difference (alpha=0.05) between the arms. To account for potential dropout, we will seek to enroll 130 patients total, 65 in each arm.

#### **Funding:**

We have applied for an IRMF grant.

## **Copying Data Already Collected:**

Some of the questionnaires for this study are the same as the questionnaires for the study Family Presence (IRB #1050086). To avoid asking subjects the same questions multiple times in a short time period, if subjects have consented to this study and were previously consented and enrolled in the other study, responses to the same questionnaires in the other study will be copied into the data for this study.

#### References:

- 1. McKiernan M, McCarthy G. Family members' lived experience in the intensive care unit: a phemenological study. *Intensive Crit. Care Nurs.* 2010;26(5):254-261.
- 2. Anderson WG, Arnold RM, Angus DC, Bryce CL. Posttraumatic stress and complicated grief in family members of patients in the intensive care unit. *J. Gen. Intern. Med.* 2008;23(11):1871-1876.
- 3. Azoulay E, Pochard F, Kentish-Barnes N, et al. Risk of post-traumatic stress symptoms in family members of intensive care unit patients. *Am. J. Respir. Crit. Care Med.* 2005;171(9):987-994.
- 4. Jamerson PA, Scheibmeir M, Bott MJ, Crighton F, Hinton RH, Cobb AK. The experiences of families with a relative in the intensive care unit. *Heart Lung.* 1996;25(6):467-474.
- 5. Kleiber C, Halm M, Titler M, et al. Emotional responses of family members during a critical care hospitalization. *Am. J. Crit. Care.* 1994;3(1):70-76.
- 6. Pochard F, Darmon M, Fassier T, et al. Symptoms of anxiety and depression in family members of intensive care unit patients before discharge or death. A prospective multicenter study. *J. Crit. Care.* 2005;20(1):90-96.
- 7. Wendler D, Rid A. Systematic review: the effect on surrogates of making treatment decisions for others. *Ann. Intern. Med.* 2011;154(5):336-346.
- 8. Netzer G, Sullivan DR. Recognizing, naming, and measuring a family intensive care unit syndrome. *Ann Am Thorac Soc.* 2014;11(3):435-441.
- 9. Cassell EJ, Leon AC, Kaufman SG. Preliminary evidence of impaired thinking in sick patients. *Ann. Intern. Med.* 2001;134(12):1120-1123.
- 10. Needham DM, Davidson J, Cohen H, et al. Improving long-term outcomes after discharge from intensive care unit: report from a stakeholders' conference. *Critical care medicine*. 2012;40(2):502-509.
- 11. Tedeschi RC, LG. *Trauma and transformation: Growing in the aftermath of suffering.* Thousand Oaks, CA: Sage Publications, Inc; 1995.
- 12. Janoff-Bulman R. *Shattered assumptions: Towards a new psychology of trauma.* New York: Free Press; 1992.
- 13. Joseph S, Linley PA. Growth following adversity: theoretical perspectives and implications for clinical practice. *Clin. Psychol. Rev.* 2006;26(8):1041-1053.
- 14. Dekel S, Mandl C, Solomon Z. Shared and unique predictors of post-traumatic growth and distress. *J. Clin. Psychol.* 2011;67(3):241-252.
- 15. Linley PA, Joseph S. Positive change following trauma and adversity: a review. *J. Trauma. Stress.* 2004;17(1):11-21.
- 16. Ogińska-Bulik N. The role of social support in posttraumatic growth in people struggling with cancer. *Health Psychology Report*. 2013;1(1):1-8.
- 17. Swickert R, Hittner J. Social support coping mediates the relationship between gender and posttraumatic growth. *J. Health Psychol.* 2009;14(3):387-393.
- 18. Frazier P, Conlon A, Glaser T. Positive and negative life changes following sexual assault. *J. Consult. Clin. Psychol.* 2001;69(6):1048-1055.
- 19. McMillen JC, Smith EM, Fisher RH. Perceived benefit and mental health after three types of disaster. *J. Consult. Clin. Psychol.* 1997;65(5):733-739.

- 20. Affleck G, Tennen H, Croog S, Levine S. Causal attribution, perceived benefits, and morbidity after a heart attack: an 8-year study. *J. Consult. Clin. Psychol.* 1987;55(1):29-35.
- 21. Pennebaker JW, Beall SK. Confronting a traumatic event: toward an understanding of inhibition and disease. *J. Abnorm. Psychol.* 1986;95(3):274-281.
- 22. Danoff-Burg SA, JD; Romanoff, NR; Kremer, JM; Strosberg, JM. Benefit finding and expressive writing in adults with lupus or rheumatoid arthritis. *Psychology and Health*. 2006;21(5):651-665.
- 23. Stockton H, Joseph, S, Hunt, N. Expressive writing and posttraumatic growth: An internet-based study. *Traumatology: An International Journal*. 2014;20(2):75-83.
- 24. Low CA, Stanton AL, Danoff-Burg S. Expressive disclosure and benefit finding among breast cancer patients: mechanisms for positive health effects. *Health Psychol.* 2006;25(2):181-189.
- 25. Koopman C, Ismailji T, Holmes D, Classen CC, Palesh O, Wales T. The effects of expressive writing on pain, depression and posttraumatic stress disorder symptoms in survivors of intimate partner violence. *J. Health Psychol.* 2005;10(2):211-221.
- 26. DiGangi JA, Gomez D, Mendoza L, Jason LA, Keys CB, Koenen KC. Pretrauma risk factors for posttraumatic stress disorder: a systematic review of the literature. *Clin. Psychol. Rev.* 2013;33(6):728-744.
- 27. Khalaila R. Patients' family satisfaction with needs met at the medical intensive care unit. *J. Adv. Nurs.* 2013;69(5):1172-1182.
- 28. Lautrette A, Darmon M, Megarbane B, et al. A communication strategy and brochure for relatives of patients dying in the ICU. *N. Engl. J. Med.* 2007;356(5):469-478.
- 29. Butler J, Hirshberg EL, Hopkins RO, et al. Preliminary identification of coping profiles relevant to surrogate decision making in the ICU. *PLoS One*. (Under review).
- 30. Adam EK, Kumari M. Assessing salivary cortisol in large-scale, epidemiological research. *Psychoneuroendocrinology.* 2009;34(10):1423-1436.
- 31. Therrien F, Drapeau V, Lalonde J, et al. Awakening cortisol response in lean, obese, and reduced obese individuals: effect of gender and fat distribution. *Obesity (Silver Spring, Md.)*. 2007;15(2):377- 385.
- 32. Butler JM, Hirshberg EL, Hopkins RO, et al. Identification of intensive care unit preferences and attributes clusters and stimulated family decision making in critical illness. *BMJ: Supportive & Pallitive Care.* 2015.
- 33. Ware JE, Jr., Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. *Med. Care.* 1992;30(6):473-483.
- 34. Bienvenu OJ, Williams JB, Yang A, Hopkins RO, Needham DM. Posttraumatic stress disorder in survivors of acute lung injury: evaluating the Impact of Event Scale-Revised. *Chest*. 2013;144(1):24-31.
- 35. Weiss DS, Marmar CR. The impact of event scale-revised. *Assessing Psychological Trauma and PTSD*. 2004;2:168-189.
- 36. Cohen S, Williamson G. Perceived Stress in a Probability Sample of the United States. In: Spacapan S, Oskamp S, eds. *The Social Psychology of Health*. Newbury Park, CA: Sage; 1988:31-67.
- 37. Cohen S, Janicki-Deverts D. Who's Stressed? Distributions of psychological stress in the United States in probability samples from 1983, 2006 and 2009. *J. Appl. Soc. Psychol.* 2012;42:1320-1334.

- 38. Carver CS. You want to measure coping but your protocol's too long: consider the brief COPE. *Int. J. Behav. Med.* 1997;4(1):92-100.
- 39. Rammstedt B, & John, O.P. . Measuring personality in one minute or less: A 10-item short version of the Big Five Inventory in English and German. . *Journal of Research in Personality*. 2007;41:203-212.
- 40. Choi J, Hoffman LA, Schulz R, et al. Health risk behaviors in family caregivers during patients' stay in intensive care units: a pilot analysis. *Am. J. Crit. Care.* 2013;22(1):41-45.
- 41. Choi J, Hoffman LA, Schulz R, et al. Self-reported physical symptoms in intensive care unit (ICU) survivors: pilot exploration over four months post-ICU discharge. *J. Pain Symptom Manage*. 2014;47(2):257-270.
- 42. Choi J, Sherwood PR, Schulz R, et al. Patterns of depressive symptoms in caregivers of mechanically ventilated critically ill adults from intensive care unit admission to 2 months postintensive care unit discharge: a pilot study. *Crit. Care Med.* 2012;40(5):1546-1553.
- 43. Bedard M, Molloy DW, Squire L, Dubois S, Lever JA, O'Donnell M. The Zarit Burden Interview: a new short version and screening version. *Gerontologist*. 2001;41(5):652-657.
- 44. Zarit SH, Orr NK, Zarit JM. *The hidden victims of Alzheimer's disease: Families under stress.* New York: New York University Press; 1985.
- 45. Zarit SH, Reever KE, Bach-Peterson J. Relatives of the impaired elderly: correlates of feelings of burden. *Gerontologist*. 1980;20(6):649-655.
- 46. Im K, Belle SH, Schulz R, Mendelsohn AB, Chelluri L. Prevalence and outcomes of caregiving after prolonged (> or =48 hours) mechanical ventilation in the ICU. *Chest.* 2004;125(2):597-606.
- 47. Williamson GM, Schulz R. Pain, activity restriction, and symptoms of depression among community- residing elderly adults. *J. Gerontol.* 1992;47(6):P367-372.
- 48. Van Pelt DC, Milbrandt EB, Qin L, et al. Informal caregiver burden among survivors of prolonged mechanical ventilation. *Am. J. Respir. Crit. Care Med.* 2007;175(2):167-173.
- 49. Van Pelt DC, Schulz R, Chelluri L, Pinsky MR. Patient-specific, time-varying predictors of post-ICU informal caregiver burden: the caregiver outcomes after ICU discharge project. *Chest.* 2010;137(1):88-94.
- 50. Greenberg MA, Stone AA. Emotional disclosure about traumas and its relation to health: effects of previous disclosure and trauma severity. *J. Pers. Soc. Psychol.* 1992;63(1):75-84.
- 51. Tedeschi RG, Calhoun LG. The Posttraumatic Growth Inventory: measuring the positive legacy of trauma. *J. Trauma. Stress.* 1996;9(3):455-471.
- 52. Pollard C, Kennedy P. A longitudinal analysis of emotional impact, coping strategies and post-traumatic psychological growth following spinal cord injury: a 10-year review. *Br. J. Health Psychol.* 2007;12(Pt 3):347-362.
- 53. Morrill EF, Brewer NT, O'Neill SC, et al. The interaction of post-traumatic growth and post-traumatic stress symptoms in predicting depressive symptoms and quality of life. *Psychooncology*. 2008;17(9):948-953.
- 54. Calhoun LG, Cann A, Tedeschi RG, McMillan J. A correlational test of the relationship between posttraumatic growth, religion, and cognitive processing. *J. Trauma. Stress.* 2000;13(3):521-527.
- 55. Kashdan TB, Kane JQ. Posttraumatic distress and the presence of posttraumatic growth and meaning in life: Experiential avoidance as a moderator. *Pers. Individ. Dif.* 2011;50(1):84-89.

# **Appendixes:**

Include survey tools, data collection forms, etc.

- Appendix 1. (IESR, HADS, and Brief Cope)
- **Appendix 2. Post Traumatic Growth Inventory**
- **Appendix 3. Essay Evaluation Measure**
- **Appendix 4. Groningen Activity Restriction Scale (GARS)**
- **Appendix 5. Physical Symptoms Scale**
- **Appendix 6. Social Support Index**
- **Appendix 7. Writing Instructions for ICU Experience Study Participants**

# Appendix 1. Impact of Event Scale Revised (IES-R)

Permission from Dr. Weiss by Samuel Brown, MD MS pending.

(Read the following statement to the *participant*): I really appreciate your help with these surveys. I want to ask about something else now. The following is a list of difficulties people sometimes have after stressful life events. I will read each item, and then ask you to indicate how distressing each difficulty has been for you during the <u>past 7 days</u> with respect to <u>your experience with your loved one's ICU stay</u>. How much were you distressed or bothered by these difficulties? In the questions, the word "it" refers to your experience with your loved one's ICU stay.

| | □1 Not at all |
|---|---|
| 1. Any reminder brought back feelings about it. | □₂ A little Bit |
| | □₃ Moderately |
| | □₄ Quite a bit |
| | □s Extremely |
| | □₁ Not at all |
| 2. I had trouble staying asleep. | □2 A little Bit |
| | □₃ Moderately |
| | □₄ Quite a bit |
| | ☐s Extremely |
| | □1 Not at all |
| 3. Other things kept making me think about it. | □2 A little Bit |
| | □₃ Moderately |
| | □₄ Quite a bit |
| | □s Extremely |
| | □1 Not at all |
| 4. I felt irritable and angry. | □₂ A little Bit |
| | □₃ Moderately |
| | □₄ Quite a bit |
| | □s Extremely |
| | □1 Not at all |
| 5. I avoided letting myself get upset when I thought about it or was | □₂ A little Bit |
| reminded of it. | □₃ Moderately |
| | □4 Quite a bit |
| | □s Extremely |
| | □1 Not at all |
| 6. I thought about it when I didn't mean to. | □₂ A little Bit |
| | □₃ Moderately |
| | □₄ Quite a bit |
| | □s Extremely |
| | □1 Not at all |
| 7. I felt as if it hadn't happened or wasn't real. | □₂ A little Bit |
| | □₃ Moderately |
| | □₄ Quite a bit |
| | Πε Extremely |

| 8. I stayed away from reminders of it. | □1 Not at all □2 A little Bit |
|---|---|
| | □₃ Moderately |
| | □4 Quite a bit |
| | □s Extremely |
| | □₁ Not at all |
| 9. Pictures about it popped into my mind. | □₂ A little Bit |
| , | □₃ Moderately |
| | □4 Quite a bit |
| | □s Extremely |
| | □₁ Not at all |
| 10. I was jumpy and easily startled. | □2 A little Bit |
| 10.1 was jumpy and easily startied. | ☐3 Moderately |
| | - |
| | □4 Quite a bit |
| | □₅Extremely |
| | □1 Not at all |
| 11. I tried not to think about it. | □₂ A little Bit |
| | □₃ Moderately |
| | □₄ Quite a bit |
| | □s Extremely |
| | □₁ Not at all |
| 12. I was aware that I still had a lot of feelings about it, but I didn't | □₂ A little Bit |
| deal with them. | □₃ Moderately |
| | □4 Quite a bit |
| | □s Extremely |
| | □₁ Not at all |
| 13. My feelings about it were kind of numb. | □2 A little Bit |
| 13. Wy recinigs about it were kind of namb. | ☐3 Moderately |
| | □4 Quite a bit |
| | □s Extremely |
| 44 I found association and alternative to the state of th | □1 Not at all |
| 14. I found myself acting or feeling like I was back at that time. | □₂ A little Bit |
| | □₃ Moderately |
| | □₄ Quite a bit |
| | □s Extremely |
| | □1 Not at all |
| 15. I had trouble falling asleep. | □₂ A little Bit |
| | □₃ Moderately |
| | □₄ Quite a bit |
| | □s Extremely |
| | □1 Not at all |
| 16. I had waves of strong feelings about it. | □₂ A little Bit |
| | □₃ Moderately |
| | □₄ Quite a bit |
| | □s Extremely |
| | □₁ Not at all |
| 17. I tried to remove it from my memory. | □2 A little Bit |
| | ☐₃ Moderately |
| | □4 Quite a bit |
| | ☐ ☐ Extremely |

| | □1 Not at all |
|---|---|
| 18. I had trouble concentrating. | □₂ A little Bit |
| | □₃ Moderately |
| | □4 Quite a bit |
| | □ <sub>5</sub> Extremely |
| | □₁ Not at all |
| 19. Reminders of it caused me to have physical reactions, such as sweating, | □₂ A little Bit |
| trouble breathing, nausea, or a pounding heart. | □₃ Moderately |
| | □₄ Quite a bit |
| | □ <sub>5</sub> Extremely |
| | □₁ Not at all |
| 20. I had dreams about it. | □₂ A little Bit |
| | □₃ Moderately |
| | □4 Quite a bit |
| | □ <sub>5</sub> Extremely |
| | □1 Not at all |
| 21. I felt watchful and on guard. | □2 A little Bit |
| | □₃ Moderately |
| | □4 Quite a bit |
| | □s Extremely |
| | □1 Not at all |
| 22. I tried not to talk about it. | □₂ A little Bit |
| | □₃ Moderately |
| | □₄ Quite a bit |
| | □s Extremely |

# Hospital Anxiety and Depression Scale (HADS) License from GL Assessment pending.

Record responses directly on licensed copy of instrument from Nfer Nelson, UK & include with CRF

(Read the following introduction to the participant): I am now going to ask some different questions. Doctors are aware that emotions play an important part in most illnesses. This questionnaire is designed to help us to know how you feel. I will read each item with the possible responses. Please respond with the reply that comes closest to how you have been feeling in the past week. Don't take too long over your replies: your immediate reaction to each item will probably be more accurate than a long, thought out response.

| 1. | I feel tense or 'wound up' | $\square_1$ Most of the time |
|---|---|---|
| | | □₂ A lot of the time |
| | | ☐₃ From time to time, occasionally |
| | | □₄ Not at all |
| 2. | I still enjoy the things I used to enjoy | □₁ Definitely as much |
| | | □₂ Not quite so much |
| | | □₃ Only a little |
| | | □4 Hardly at all |
| 3. | I get a sort of frightened feeling as if | □1 Very definitely and quite badly |
| | something awful is about to happen | □₂ Yes, but not too badly |
| | | □₃ A little, but it doesn't worry me |
| | | □₄ Not at all |
| 4 | | |
| 4. | I can laugh and see the funny side of things | $\square_1$ As much as I always could |
| 4. | i can laugh and see the funny side of things | □ As much as I always could □ Not quite so much now |
| 4. | i can laugh and see the funny side of things | · |
| 4. | i can laugh and see the funny side of things | □₂ Not quite so much now |
| 5. | Worrying thoughts go through my mind | ☐2 Not quite so much now ☐3 Definitely not so much now |
| | | ☐2 Not quite so much now ☐3 Definitely not so much now ☐4 Not at all |
| | | □² Not quite so much now □³ Definitely not so much now □⁴ Not at all □¹ A great deal of the time |
| | | □² Not quite so much now □³ Definitely not so much now □⁴ Not at all □¹ A great deal of the time □² A lot of the time |
| | | □² Not quite so much now □³ Definitely not so much now □⁴ Not at all □¹ A great deal of the time □² A lot of the time □³ From time to time but not too often |
| 5. | Worrying thoughts go through my mind | □² Not quite so much now □³ Definitely not so much now □⁴ Not at all □¹ A great deal of the time □² A lot of the time □³ From time to time but not too often □⁴ Only occasionally |
| 5. | Worrying thoughts go through my mind | □² Not quite so much now □³ Definitely not so much now □⁴ Not at all □¹ A great deal of the time □² A lot of the time □³ From time to time but not too often □⁴ Only occasionally □¹ Not at all |

| 7. I can sit at ease and feel relaxed | □1 Not at all |
|---|---|
| | □₂ Not often |
| | □₃ Sometimes |
| | □4 Most of the time |
| 8. I feel as if I am slowed down | □1 Nearly all the time |
| | □₂ Very often |
| | □₃ Sometimes |
| | □4 Not at all |
| 9. I get a sort of frightened feeling like 'butterflies' | □1 Not at all |
| in the stomach | □2 Occasionally |
| | □₃ Quite often |
| | □4 Very often |
| 10. I have lost interest in my appearance | □1 Definitely |
| | □2 I don't take so much care as I should |
| | □₃ I may not take quite as much care |
| | □41 take just as much care as ever |
| 11. I feel restless, as if I have to be on the move | □₁ Very much indeed |
| | □₂ Quite a lot |
| | □ <sub>3</sub> Not very much |
| | □4 Not at all |
| 12. I look forward with enjoyment to things | □1 As much as I ever did |
| | □₂ Rather less than I used to |
| | □₃ Definitely less than I used to |
| | □4 Hardly at all |
| 13. I get sudden feelings of panic | □1 Very often indeed |
| | □₂ Quite often |
| | □₃ Not very often |
| | □4 Not at all |
| 14. I can enjoy a good book or radio or TV program | □1 Often |
| | □₂ Sometimes |
| | □₃ Not often |
| | □4 Very Seldom |

# **Coping with Stress (Brief COPE)**

| | I haven't<br>been doing<br>this at all | I've been<br>doing this a<br>little bit | I've been<br>doing this a<br>medium<br>amount | I've been doing<br>this a lot |
|---|---|---|---|---|
| 1. I've been turning to work or other activities to take my mind off of things | 1 | 2 | 3 | 4 |
| 2. I've been concentrating my efforts on doing something about the situation I'm in. | 1 | 2 | 3 | 4 |
| 3. I've been saying to myself "this isn't real.". | 1 | 2 | 3 | 4 |
| 4. I've been using alcohol or other drugs to make myself feel better. | 1 | 2 | 3 | 4 |
| 5. I've been getting emotional support from others. | 1 | 2 | 3 | 4 |
| 6. I've been giving up trying to deal with it. | 1 | 2 | 3 | 4 |
| 7. I've been taking action to try to make the situation better. | 1 | 2 | 3 | 4 |
| 8. I've been refusing to believe that it has happened. | 1 | 2 | 3 | 4 |
| 9. I've been saying things to let my unpleasant feelings escape. | 1 | 2 | 3 | 4 |
| 10. I've been getting help and advice from other people. | 1 | 2 | 3 | 4 |
| 11. I've been using alcohol or other drugs to help me get through it. | 1 | 2 | 3 | 4 |
| 12. I've been trying to see it in a different light, to make it seem more positive. | 1 | 2 | 3 | 4 |
| 13. I've been criticizing myself. | 1 | 2 | 3 | 4 |
| 14. I've been trying to come up with a strategy about what to do. | 1 | 2 | 3 | 4 |
| 15. I've been getting comfort and understanding from someone. | 1 | 2 | 3 | 4 |
| 16. I've been giving up the attempt to cope. | 1 | 2 | 3 | 4 |
| 17. I've been looking for something good in what is happening. | 1 | 2 | 3 | 4 |
| 18. I've been making jokes about it. | 1 | 2 | 3 | 4 |
| 19. I've been doing something to think about it less, such as going to movies, watching TV, reading, daydreaming, sleeping, or shopping. | 1 | 2 | 3 | 4 |

20. I've been accepting the reality of the fact that it has happened. 21. I've been expressing my negative feelings. 22. I've been trying to find comfort in my religion or spiritual beliefs. 23. I've been trying to get advice or help from other people about what to do. 24. I've been learning to live with it. 25. I've been thinking hard about what steps to take. 26. I've been blaming myself for things that happened. 27. I've been praying or meditating 28. I've been making fun of the situation 

# **Appendix 2. Post Traumatic Growth Inventory**

**Instructions**: Please indicate for each of the statements below the degree to which this change occurred in your life as a result of your crisis, using the following scale.

| | I did not | 1 | 1 | 1 | I | I |
|---|---|---|---|---|---|---|
| | experience | experienced | experienced | experienced | experienced | experienced |
| | this | this change | this change | this change | this change | this change |
| | change as | to a very | to a small | to a | to a great | to a very |
| | a result of | small degree | degree as a | moderate | degree as a | great degree |
| | my crisis | as a result of | result of my | degree as a | result of my | as a result of |
| | | my crisis | crisis | result of my | crisis | my crisis |
| My priorities | | | | | | |
| about what is | 0 | 1 | 2 | 3 | 4 | 5 |
| important in life | | | | | | |
| An appreciation | | | | | | |
| for the value of | 0 | 1 | 2 | 3 | 4 | 5 |
| my own life | | | | | | |
| I developed new | | | | | | |
| interests | 0 | 1 | 2 | 3 | 4 | 5 |
| A feeling of self- | | _ | | | _ | _ |
| reliance | 0 | 1 | 2 | 3 | 4 | 5 |
| A better | | | | | | |
| understanding of | 0 | 1 | 2 | 3 | 4 | 5 |
| spiritual matters | | | | | | |
| Knowing that I | | | | | | |
| can count on | 0 | 1 | 2 | 3 | 4 | 5 |
| people in times | | | | | | |
| of trouble | | | | | | |
| I established a | | | | | | |
| new path for my | 0 | 1 | 2 | 3 | 4 | 5 |
| life | | | | | | |
| A sense of | | | | | | |
| closeness with | 0 | 1 | 2 | 3 | 4 | 5 |
| others | | | | | | |
| A willingness to | | | | | | |
| express my | 0 | 1 | 2 | 3 | 4 | 5 |
| emotions | | | | | | |
| Knowing I can | | | | | | |
| handle | 0 | 1 | 2 | 3 | 4 | 5 |
| difficulties | | | | | | |
| I'm able to do | | | | | | |
| better things | 0 | 1 | 2 | 3 | 4 | 5 |
| with my life | | | | | | |

| | 1 | 1 | I | | | |
|---|---|---|---|---|---|---|
| | I did not | I | I | I | I | I |
| | experience | experienced | experienced | experienced | experienced | experienced |
| | this | this change | this change | this change | this change | this change |
| | change as | to a very | to a small | to a | to a great | to a very |
| | a result of | small degree | degree as a | moderate | degree as a | great degree |
| | my crisis | as a result of | result of my | degree as a | result of my | as a result of |
| | , | my crisis | crisis | result of my | crisis | my crisis |
| Being able to | | , | | , | | , |
| accept the way | 0 | 1 | 2 | 3 | 4 | 5 |
| things work out | | _ | _ | | | |
| Appreciating | | | | | | |
| each day | 0 | 1 | 2 | 3 | 4 | 5 |
| eachiday | U | 1 | 2 | 3 | 4 | 5 |
| New | | | | | | |
| opportunities | 0 | 1 | 2 | 3 | 4 | 5 |
| are available | | _ | _ | | - | |
| which | | | | | | |
| wouldn't have | | | | | | |
| been | | | | | | |
| Having | 0 | 1 | 2 | 3 | 4 | 5 |
| compassion for | 0 | 1 | 2 | 3 | 4 | 5 |
| others | | | | | | |
| Putting effort | | | | | | |
| _ | | 1 | 2 | 3 | 4 | 5 |
| into my | 0 | 1 | | 3 | 4 | 5 |
| relationships | | | | | | |
| I'm more likely | | | | | _ | _ |
| to try to change | 0 | 1 | 2 | 3 | 4 | 5 |
| things which | | | | | | |
| need changing | | | | | | |
| I have a | | | | | | |
| stronger | 0 | 1 | 2 | 3 | 4 | 5 |
| religious faith | | | | | | |
| I discovered | | | | | | |
| that I'm | 0 | 1 | 2 | 3 | 4 | 5 |
| stronger than I | | | | | | |
| thought I was | | | | | | |
| I learned a great | | | | | | |
| deal about how | 0 | 1 | 2 | 3 | 4 | 5 |
| wonderful | | _ | _ | | | |
| people are | | | | | | |
| I accept needing | | | | | | |
| others | 0 | 1 | 2 | 3 | 4 | 5 |
| Others | | | _ | | 7 | , |
| | 1 | | | | | |

# **Appendix 3. Essay Evaluation Measure**

**Instructions**: Please answer the following questions about your essay using the scale provided.

| | Not at<br>All | Low | Slightly | Neutral | Moderately | Very | A Great<br>Deal |
|---|---|---|---|---|---|---|---|
| How personal was the essay that you wrote today? | 0 | 1 | 2 | 3 | 4 | 5 | 6 |
| How much did you reveal your emotions in what you wrote today? | 0 | 1 | 2 | 3 | 4 | 5 | 6 |
| Have much of what you wrote today have you shared with/told others? | 0 | 1 | 2 | 3 | 4 | 5 | 6 |

# Appendix 4.

# **Groningen Activity Restriction Scale (GARS)**

The following questions refer to daily activit ies which should be performed frequently. In each question it is asked whether you are able to perform the activity at this moment. It is not intended to assess whether you are actually performing the activities, but if you can do them if necessary. Response categories for each item

- 1. Yes, I can do it fully independently without any difficulty
- 2. Yes, I can do it fully independently but with some difficulty
- 3. Yes, I can do it fully independently but with great difficulty
- 4. No, I cannot do it fully independently, I can only do it with someone's help GARS items
- 1. Can you, fully independently, dress yourself?
- 2. Can you, fully independently, get in and out of bed?
- 3. Can you, fully independently, stand up from sitting in a chair?
- 4. Can you, fully independently, wash your face and hands?
- 5. Can you, fully independently, wash and dry your whole body?
- 6. Can you, fully independently, get on and off the toilet?
- 7. Can you, fully independently, feed yourself?
- 8. Can you, fully independently, get around in the house (if necessary with a cane or walker)?
- 9. Can you, fully independently, go up and down the stairs?
- 10. Can you, fully independently, walk outdoors (if necessary with a cane or walker)?
- 11. Can you, fully independently, take care of your feet and toenails?
- 12. Can you, fully independently, prepare breakfast or lunch?
- 13. Can you, fully independently, prepare dinner?
- 14. Can you, fully independently, do "light" household activities (for example, dusting and tidying up)?
- 15. Can you, fully independently, do "heavy" household activities (for example mopping, cleaning the windows, and vacuuming)?
- 16. Can you, fully independently, wash and iron your clothes?
- 17. Can you, fully independently, make the beds?
- 18. Can you, fully independently, do the shopping?

## **Activity Restriction Scale (ARS)**

| "Please tell me how much you have restricted your activities in each of the following areas due to the | |
|---|---|
| care you are providing to your loved one: | |
| 1. Care of yourself? | □₁ Not restricted at all |
| | □ <sub>2</sub> Slightly restricted |
| | □₃ Moderately restricted |
| | □ <sub>4</sub> Greatly restricted |
| 2. Caring for others? | □1 Not restricted at all |
| | □ <sub>2</sub> Slightly restricted |
| | □₃ Moderately restricted |
| | □4 Greatly restricted |

| 3. | Eating habits? | □₁ Not restricted at all |
|---|---|---|
| J. | Lating nabits: | |
| | | □2 Slightly restricted |
| | | □ <sub>3</sub> Moderately restricted |
| 4 | Classing habita? | □4 Greatly restricted |
| 4. | Sleeping habits? | □1 Not restricted at all |
| | | □2 Slightly restricted |
| | | □ <sub>3</sub> Moderately restricted |
| - | D: 1 111 2 | □4 Greatly restricted |
| 5. | Doing household chores? | □¹ Not restricted at all |
| | | □2 Slightly restricted |
| | | □ <sub>3</sub> Moderately restricted |
| - | | □ 4 Greatly restricted |
| 6. | Going shopping for him/herself | □1 Not restricted at all |
| | | □2 Slightly restricted |
| | | □ <sub>3</sub> Moderately restricted |
| | | □4 Greatly restricted |
| 7. | Visiting friends? | □¹ Not restricted at all |
| | | □ <sub>2</sub> Slightly restricted |
| | | □ <sub>3</sub> Moderately restricted |
| | | □4 Greatly restricted |
| 8. | Working on hobbies? | □1 Not restricted at all |
| | | □ <sub>2</sub> Slightly restricted |
| | | □₃ Moderately restricted |
| | | □4 Greatly restricted |
| 9. | Sports and recreation? | □1 Not restricted at all |
| | | □ <sub>2</sub> Slightly restricted |
| | | □₃ Moderately restricted |
| | | □4 Greatly restricted |
| 10. | Going to work? | □₁ Not restricted at all |
| | | □ <sub>2</sub> Slightly restricted |
| | | □₃ Moderately restricted |
| | | □4 Greatly restricted |
| 11. | Maintaining friendship? | □1 Not restricted at all |
| _ <del></del> | | □2 Slightly restricted |
| | | □₃ Moderately restricted |
| | | □4 Greatly restricted |
| | | Li4 Greatly restricted |

# **Appendix 5. Physical Symptoms Scale**

**Instructions**: On how many of the past 30 days have you experienced each of the following symptoms?

| | Number of Days |
|-------------------------|----------------|
| | 0-30 |
| Headache | |
| Stomach Ache/Pain/Upset | |
| Chest Pain | |
| Runny/Congested Nose | |
| Coughing/Sore Throat | |
| Faintness/Dizziness | |
| Shortness of Breath | |
| Racing/Pounding Heart | |
| Stiff/Sore Muscles | |

**Instructions**: In the past 30 days, have you seen a doctor/health care professional for treatment for any of these symptoms?

| | Yes | No |
|-------------------------|-----|----|
| Headache | | |
| Stomach Ache/Pain/Upset | | |
| Chest Pain | | |
| Runny/Congested Nose | | |
| Coughing/Sore Throat | | |
| Faintness/Dizziness | | |
| Shortness of Breath | | |
| Racing/Pounding Heart | | |
| Stiff/Sore Muscles | | |

# **Appendix 6. Social Support**

**Instructions:** When we need support such as advice, understanding or a favor, our relationship with other people (for example, parents, spouses, friends), may or may not have both helpful and upsetting aspects. For the person **most important** to you, please complete the following.

- Specify the relationship to you (such as a spouse, sister, co-worker, or friend) and the gender of the person
- Provide an estimate of the length of time you have known this person, and the average number
  of times per week you have contact with this person
- When you need support such as advice, understanding or a favor, rate this person on:
  - o How generally helpful this person is to you (using the scale titled "HOW HELPFUL?")
  - How generally upsetting this person is to you (using the scale titled "HOW UPSETTING?")

(Note: When asked to rate the extent the individual is HELPFUL, you should ignore any upsetting aspects of the relationship. When asked to rate the extent the individual is UPSETTING, you should ignore any helpful aspects of the relationship.)

• For the final rating, indicate how unpredictable the person is when you need support such as advice, understanding or a favor.

| Initials of person most Important to you. | Relationship<br>to you. | Gender<br>of<br>person. | Appropriate length of time you have known the person (years or months). | Average number of times per week you have contact with the person. | HOW HELPFUL is this person to you? 1 = Not at all helpful 2 = A little helpful 3 = Somewhat helpful 4 = Moderately helpful 5 = Very helpful 6 = Extremely helpful (Circle one number) | HOW UPSETTING is this person to you? 1 = Not at all upsetting 2 = A little upsetting 3 = Somewhat upsetting 4 = Moderately upsetting 5 = Very upsetting 6 = Extremely upsetting (Circle one | HOW UNPREDICTABLE is this person to you? 1 = Not at all unpredictable 2 = A little unpredictable 3 = Somewhat unpredictable 4 = Moderately unpredictable 5 = Very unpredictable 6 = Extremely unpredictable (Circle one number) |
|---|---|---|---|---|---|---|---|
| | | | | | 123456 | number)<br>1 2 3 4 5 6 | 123456 |

# Appendix 7. Writing Instructions for ICU Experience Study Participants

# Writing Instructions for Study Participants (A)

Thank you for agreeing to complete the writing part of this study at home. Below are instructions for the writing session.

- 1. You have been assigned a unique identifier to use instead of your name. For example, your identifier could be **193JAO**.
- 2. Writing session: You will write for 20 minutes on your computer, take a 10 to 15-minute break and then write for 20 minutes. After the second writing sessions take a 10 to 15-minute break and write for 20 minutes (third writing session).
- 3. Save each writing session to your computer, please save your writing. Title the document as the unique identifier (193JAO) we sent you and ICU Experience. Example: 193JAO ICU Experience. Save the writing to your computer.
- 4. Label each writing session. The first one should be writing 1. The second writing as writing 2 and the third as writing 3. All three writing sessions can be saved in one document, but please label each one so we know which session is which (session 1, session 2, or session 3).
- 5. Prior to starting each writing session, please read the instructions below.

#### **Writing Instructions**

"What I would like you to write about for these three sessions are your deepest thoughts and feelings about your experience with your family member in the Intensive Care Unit (ICU). I realize that people with a loved one in the ICU experience a full range of emotions and thoughts, and I want you to focus on any and all of them. In your writing, I want you to really let go and explore your very deepest emotions and thoughts. You might think about all the various feelings and changes that you experienced before your loved one was hospitalized in the ICU, after the diagnosis that led them to the ICU, during treatment, and now. Whatever you choose to write, it is critical that you really focus on your deepest thoughts and feelings. Ideally, I would like you to focus on feelings, thoughts, or changes that you have not discussed in great detail with others- private feelings. You might also tie your thoughts and feelings about your experiences with having your loved one in the ICU to other parts of your life, i.e., your childhood, people you love (this loved one and others), who you are, or who you want to be. Again, the most important part of your writing is that you really focus on your deepest emotions and thoughts. The only rule we have is that you write continuously for the entire time. If you run out of things to say, just repeat what you have already written. Don't worry about grammar, spelling, or sentence structure. Don't worry about erasing or crossing things out. Just write."

6. Once you have completed your writing, email your writing to Mardee Merrill at <a href="Mardee.Merrill@imail.org">Mardee.Merrill@imail.org</a> or to Ramona Hopkins, PhD at <a href="Mona.Hopkins@imail.org">Mona.Hopkins@imail.org</a>. In the subject line put your identifier, in this example 193JAO.

Please contact Mardee Merrill if you have any questions at 801-507-4608 or Mardee.Merril@imail.org.

# Writing Instructions for Study Participants (B)

Thank you for agreeing to complete the writing part of this study at home. Below are instructions for the writing session.

- 1. You have been assigned a unique identifier to use instead of your name. For example, your identifier could be **193JAO**.
- 2. Writing session: You will write for 20 minutes, take a 10 to 15-minute break and then write for 20 minutes. After the second writing sessions take a 10 to 15-minute break and write for 20 minutes (third writing session).
- 3. Save each writing session to your computer, please save your writing. Title the document as the unique identifier (193JAO) we sent you and ICU Experience. Example: 193JAO ICU Experience. Save the writing to your computer.
- 4. Label each writing session The first one should be writing 1. The second writing as writing 2 and the third as writing 3. All three writing sessions can be saved in one document, but please label each one so we know which session is which (session 1, session 2, or session 3).
- 5. Prior to starting each writing session, please read the instructions below.

"What I would like you to write about for these three sessions are all the facts about your experience with your family member in the Intensive Care Unit (ICU). We are not interested in your thoughts and emotions. Please do not include them. We are interested in all the facts about how your loved one came to the ICU and the facts about your experiences in the ICU with your loved one. The only rule we have is that you write continuously for the entire time. If you run out of things to say, just repeat what you have already written. Don't worry about grammar, spelling, or sentence structure. Don't worry about erasing or crossing things out. Just write."

6. Once you have completed your writing, email your writing to Mardee Merrill at <a href="Mardee.Merrill@imail.org">Mardee.Merrill@imail.org</a> or to Ramona Hopkins, PhD at <a href="Mona.Hopkins@imail.org">Mona.Hopkins@imail.org</a>. In the subject line put your identifier, in this example 193JAO.

Please contact Mardee Merrill if you have any questions at 801-507-4608 or Mardee.Merril@imail.org.

# Writing Instructions for Study Participants who do not have a Computer (C)

Thank you for agreeing to complete the writing part of this study at home. Below are instructions for the writing session.

1. You have been assigned a unique identifier to use instead of your name. For example, your identifier could be **193JAO**.

2. Writing session: You will write for 20 minutes long-hand, take a 10 to 15-minute break and then write for 20 minutes. After the second writing sessions take a 10 to 15-minute break and write for 20 minutes (third writing session).

- 3. Title the document as the unique identifier (193JAO) we sent you and staple together if possible.
- 4. Label each writing session. The first one should be writing 1. The second writing as writing 2 and the third as writing 3. All three can be in one document, but please label each writing session so we can tell which is which.
- 5. Prior to starting each writing session, please read the instructions below.

## **Writing Instructions**

"What I would like you to write about for these three sessions are your deepest thoughts and feelings about your experience with your family member in the Intensive Care Unit (ICU). I realize that people with a loved one in the ICU experience a full range of emotions and thoughts, and I want you to focus on any and all of them. In your writing, I want you to really let go and explore your very deepest emotions and thoughts. You might think about all the various feelings and changes that you experienced before your loved one was hospitalized in the ICU, after the diagnosis that led them to the ICU, during treatment, and now. Whatever you choose to write, it is critical that you really focus on your deepest thoughts and feelings. Ideally, I would like you to focus on feelings, thoughts, or changes that you have not discussed in great detail with othersprivate feelings. You might also tie your thoughts and feelings about your experiences with having your loved one in the ICU to other parts of your life, i.e., your childhood, people you love (this loved one and others), who you are, or who you want to be. Again, the most important part of your writing is that you really focus on your deepest emotions and thoughts. The only rule we have is that you write continuously for the entire time. If you run out of things to say, just repeat what you have already written. Don't worry about grammar, spelling, or sentence structure. Don't worry about erasing or crossing things out. Just write."

6. Once you have completed your writing, you will be provided with a self-addressed stamped envelope. Please your writing sample inside and mail to:

Mardee Merrill Pulmonary Research Sorenson Heart-Lung Center, 6<sup>th</sup> floor 5121 S. Cottonwood Street Murray, Utah 84107

Please contact Mardee Merrill if you have any questions at 801-507-4608 or Mardee.Merril@imail.org.

# Writing Instructions for Study Participants who do not have a Computer (D)

Thank you for agreeing to complete the writing part of this study at home. Below are instructions for the writing session.

- 1. You have been assigned a unique identifier to use instead of your name. For example, your identifier could be **193JAO**.
- 2. Writing session: You will write for 20 minutes long-hand, take a 10 to 15-minute break and then write for 20 minutes. After the second writing sessions take a 10 to 15-minute break and write for 20 minutes (third writing session).
- 3. Title the document as the unique identifier (193JAO) we sent you and staple together if possible.
- 4. Label each writing session. The first one should be writing 1. The second writing as writing 2 and the third as writing 3. All three can be in one document, but please label each writing session so we can tell which is which.
- 5. Prior to starting each writing session, please read the instructions below.

# **Writing Instructions**

"What I would like you to write about for these three sessions are all the facts about your experience with your family member in the Intensive Care Unit (ICU). We are not interested in your thoughts and emotions. Please do not include them. We are interested in all the facts about how your loved one came to the ICU and the facts about your experiences in the ICU with your loved one. The only rule we have is that you write continuously for the entire time. If you run out of things to say, just repeat what you have already written. Don't worry about grammar, spelling, or sentence structure. Don't worry about erasing or crossing things out. Just write."

6. Once you have completed your writing, you will be provided with a self-addressed stamped envelope. Please your writing sample inside and mail to:

Mardee Merrill Pulmonary Research Sorenson Heart-Lung Center, 6<sup>th</sup> floor 5121 S. Cottonwood Street Murray, Utah 84107

Please contact Mardee Merrill if you have any questions at 801-507-4608 or Mardee.Merril@imail.org.